CLINICAL TRIAL: NCT04812886
Title: Gout in French Polynesia: Epidemiology and Comorbidities, Genetic Causes and Prevalence of HLA B58:01
Brief Title: Epidemiology of Gout in French Polynesia
Acronym: TOPATA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Variant Bio, Inc. (Unknown); University of Birmingham (Other); University of San Diego (Other); Ministry of Health, French Polynesia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC-P00104
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Gout
Keywords: Gout, French Polynesia, Epidemiology
MeSH Terms: conditions — Gout | interventions — Epidemiologic Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidemiological study (Experimental)
  Interventions: Other: Epidemiological study

INTERVENTIONS:
Other: Epidemiological study — Questionnaires (quality of life, gout, life habit, comorbidities) anthropometrics and health measures DNA analysis RNA analysis Metabolomic analysis

SUMMARY:
Gout is a chronic disease caused by the deposit of monosodium urate (MSU) crystals in body tissues secondary to hyperuricemia. Patients with gout suffer severe attacks of acute joint pain. As the disease progresses, the joint pain becomes chronic and associated with disabling and deformative manifestations called tophi. Gout is strongly associated with various comorbidities including cardiovascular disease and chronic kidney failure. Gout is a very common disease, affecting 0.9% of the adult population in France and nearly 4% of the North-American population. Data from New Zealand show a particularly high prevalence of gout among Polynesians (minority populations in New Zealand and other islands of the South Pacific) that would be explained by genetic susceptibility and frequently intertwined with metabolic diseases. Recent findings obtained from the Polynesian population in New Caledonia disclose high prevalence figures close to 7%, a level expected to be confirmed by an epidemiology study that will be conducted in parallel with the present study and designed to determine the precise prevalence of gout in French Polynesia and the most frequently associated genetic variants.

DETAILED DESCRIPTION:
International genomic studies conducted in populations with hyperuricemia and gout have identified a number of associated alleles. The strength of the association between a given allele and gout (or hyperuricemia) provides an indication of the importance of the encoded protein in disease pathogenesis. It was in this way that the development of gout was found to depend on renal urate transporters that were subsequently targeted by new uricosuric therapies.

Overall, the search for gout-associated genes has mostly been done in the general European population and revealed a small number of candidate loci. Most of these only contribute a small amount to the heritability for gout susceptibility, suggesting that additional genes and mechanisms of genetic influence are yet to be discovered. A common feature of Genome-Wide Association studies done so far is that usually large sample sizes are required in order to detect differences in allele frequencies and their contribution to different traits between test groups. The Polynesian population of French Polynesia possesses characteristics that make it particularly attractive to carry out population-based genetic research. Historical records indicate that the Polynesians of Tahiti and surrounding islands originate from a small founder population that has undergone a number of bottlenecks, eventually becoming a genetically homogenous population with a fairly high degree of consanguinity. The combination of a historic founder event, continued isolation and recent expansion are all ideal properties for a Genome Wide Association Study, as they ensure that 1) population stratification will be easy to correct when performing association tests and 2) there are likely high-effect variants that were kept at low frequency in mainland Europe due to negative selection but rose to high frequencies in the Polynesians via the increase in genetic drift or selection through adaptation to a specific environment and diet. Therefore, it is plausible that rare variants with large effect on health-related quantitative traits may be more easily detectable in Polynesians, even with much smaller sample sizes.

ELIGIBILITY:
Inclusion Criteria:

* Living in Tahiti, Moorea, Tahaa-Raiatea, Tikehau, Nuku Hiva, Mangareva, Rurutu
* Agreeing to participate in the study

Exclusion Criteria:

* Homeless
* Living in communities (military camp, hospices, university residence, ...)
* Unable to answer questionnaires
* Under guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1088 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Gout Prevalence | 6 months
  Measure of gout prevalence

SECONDARY OUTCOMES:
Diagnosis of Hyperuricemia | 6 months
  Diagnosed when uricemia is higher than 360 µmol/l
Genome wide analysis for identification of genetic variants linked to gout | 6 months
  Analysis of the genetic determinants of gout and hyperuricemia in French Polynesia via a pan-genomic analysis using complete and then rapid sequencing techniques
HLA B58:01 allele prevalence | 6 months
Multiple correlation between renal failure, diabetes, gout and cardiovascular comorbidities | 6 months
  The association between cardiovascular comorbidities/renal failure/diabetes and gout will be investigated using a multivariate logistic regression model.
Multiple correlation between renal failure, diabetes, hyperuricemia and cardiovascular comorbidities | 6 months
  The association between cardiovascular comorbidities/renal failure/diabetes and hyperuricemia will be investigated using a multivariate logistic regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Pascart, MD, PhD, Principal Investigator — GHICL
Locations (1):
- Centre Hospitalier de la Polynésie Française, Pirae, French Polynesia

IPD SHARING:
Plan to Share IPD: No